CLINICAL TRIAL: NCT05508425
Title: Comparing the Effects of Water Temperature and Actives in Glucose Solution on Pregnant Women's Taste and Side Effects During an Oral Glucose Tolerance Test-A Randomized Controlled Trial
Brief Title: Comparing the Effects of Water Temperature and Actives in Glucose Solution on Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB2021110
Record Dates: First submitted 2022-08-10; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- water at room temperature (Active Comparator)
  Interventions: Diagnostic Test: oral glucose tolerance test using water at room temperature
- hot water (Experimental)
  Interventions: Diagnostic Test: oral glucose tolerance test using hot water
- cold water (Experimental)
  Interventions: Diagnostic Test: oral glucose tolerance test using cold water
- hot water with tea bag (Experimental)
  Interventions: Diagnostic Test: oral glucose tolerance test using hot water with tea bag
- room temperature water with tea bag (Experimental)
  Interventions: Diagnostic Test: oral glucose tolerance test using room temperature water with tea bag
- cold water with tea bag (Experimental)
  Interventions: Diagnostic Test: oral glucose tolerance test using cold water with tea bag
- bubble water at room temperature (Experimental)
  Interventions: Diagnostic Test: Oral glucose tolerance test using bubble water at room temperature
- cold bubble water (Experimental)
  Interventions: Diagnostic Test: Oral glucose tolerance test using bubble water

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test using water at room temperature — The use of water at room temperature to solve the 75g glucose.
  Arms: water at room temperature
Diagnostic Test: oral glucose tolerance test using hot water — The use of hot water to solve the 75g glucose.
  Arms: hot water
Diagnostic Test: oral glucose tolerance test using cold water — The use of cold water to solve the 75g glucose.
  Arms: cold water
Diagnostic Test: oral glucose tolerance test using hot water with tea bag — The use of hot water with tea bag to solve the 75g glucose.
  Arms: hot water with tea bag
Diagnostic Test: oral glucose tolerance test using room temperature water with tea bag — The use of room temperature water with tea bag to solve the 75g glucose.
  Arms: room temperature water with tea bag
Diagnostic Test: oral glucose tolerance test using cold water with tea bag — The use of cold water with tea bag to solve the 75g glucose.
  Arms: cold water with tea bag
Diagnostic Test: Oral glucose tolerance test using bubble water at room temperature — The use of bubble water at room temperature to solve the 75g glucose.
  Arms: bubble water at room temperature
Diagnostic Test: Oral glucose tolerance test using bubble water — The use of cold bubble water to solve the 75g glucose.
  Arms: cold bubble water

SUMMARY:
To assess the effect of water temperature and additives on pregnant women's taste and side effect during the oral glucose tolerance test (OGTT) evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Gestational age between 24 and 28 weeks

Exclusion Criteria:

* Clinical diagnosis of overt type 2 diabetes
* Clinical diagnosis of facial palsy
* Clinical diagnosis of oral cavity and throat
* Clinical diagnosis of hypothyroidism
* Clinical diagnosis of chronic hepatitis
* Clinical diagnosis of kidney disease .Clinical diagnosis of Sicca syndrome.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Glycaemia level | Glycaemia level was measured just before glucose administration.
  Glycaemia level just before glucose administration
Glycaemia level | Glycaemia level was measured at 1 hour after glucose administration
  Glycaemia level at 1 hour after glucose administration
Glycaemia level | Glycaemia level was measured at 2 hours after glucose administration
  Glycaemia level at 2 hour after glucose administration
gestational diabetes mellitus | Just before glucose administration.
  gestational diabetes mellitus just before glucose administration.
gestational diabetes mellitus | At 1 hour after glucose administration
  gestational diabetes mellitus at 1 hour after glucose administration.
gestational diabetes mellitus | At 2 hour after glucose administration
  gestational diabetes mellitus at 2 hour after glucose administration.
Satisfaction after glucose solution administration | Just after glucose administration
  Satisfaction was measured by a questionnaire using 5-point Likert scale (1: very dissatisfied; 2: dissatisfied; 3: neutral; 4: satisfied; 5: very satisfied).
Taste after glucose solution administration | Just after glucose administration
  Taste was measured by a questionnaire using 5-point Likert scale (1: very dissatisfied; 2: dissatisfied; 3: neutral; 4: satisfied; 5: very satisfied).
Nausea after glucose solution administration | Just after glucose administration
  Nausea was measured by a questionnaire using 5-point Likert scale (1: not at all; 2: slightly; 3: neutral; 4: serious; 5: very serious)
Vomiting after glucose solution administration | Just after glucose solution administration
  Vomiting was measured by a questionnaire using 5-point Likert scale (1: not at all; 2: slightly; 3: neutral; 4: serious; 5: very serious)
Headache after glucose solution administration | Just after glucose solution administration
  Headache was measured by a questionnaire using 5-point Likert scale (1: not at all; 2: slightly; 3: neutral; 4: serious; 5: very serious)
Abdominal bloating after glucose solution administration | Just after glucose solution administration
  Abdominal bloating was measured by a questionnaire using 5-point Likert scale (1: not at all; 2: slightly; 3: neutral; 4: serious; 5: very serious)

CONTACTS AND LOCATIONS:
Locations (1):
- Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang P, Chang PC, Wang CY, Wang LC, Shih CL. Comparing the effects of water temperature and additives in glucose solution on pregnant women's taste, side effects, and glycemic levels during an oral glucose tolerance test: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Apr;5(4):100870. doi: 10.1016/j.ajogmf.2023.100870. Epub 2023 Jan 20. PMID 36690181